CLINICAL TRIAL: NCT01114074
Title: The Influence of the Proteins of the Contact Activation System on Thrombus Formation Under Different Flow-conditions in Blood
Brief Title: Thrombus Formation Under Different Flow-conditions
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 10-3-015; #2008B120 (Other Grant/Funding Number: Netherlands Heart Fundation)
Record Dates: First submitted 2010-04-12; First posted 2010-04-30 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Thrombosis
Keywords: Thrombosis; Blood coagulation; Perfusion flow experiments; Factor XII; Factor XI; Prekallikrein; High molecular weight kininogen
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * Whole blood
  * Platelet poor plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Factor XII deficiency: Patients deficient in coagulation factor XII
- Factor XI Deficiency: Patients deficient in coagulation factor XI
- Prekallikrein deficiency: Patients deficient in prekallikrein
- HMWK deficiency: Patients deficient in high molecular weight kininogen (HMWK)
- Control group: Healthy controls

SUMMARY:
Rationale: Cardiovascular diseases are important causes of morbidity and mortality in the industrialized world. Clinical studies indicate an important role for the proteins of the contact activation system (coagulation factor XII (FXII), FXI, prekallikrein and high molecular weight kininogen (HMWK)) on the risk of cardiovascular disease. There is substantial evidence from mouse studies that FXII and FXI participate in the formation and stability of thrombi and in vitro studies showed that collagen is able to activate FXII and hereby stimulate thrombin formation and potentiate the formation of platelet-fibrin thrombi. The investigators want to determine the role of the proteins of the contact activation system in platelet mediated thrombus formation in human blood.

Objective: The investigators will study the effects of the proteins of the contact activation system on platelet mediated thrombus formation, embolization and degradation on collagen in a perfusion flow model.

Study design: Blood will be collected from human volunteers via a venipuncture in the forearm. Each volunteer will donate maximally four times 30 ml of blood over a period of two days. This blood is used in perfusion flow experiments: blood flows over a coverslip covered with collagen in a flow chamber. The investigators will vary several conditions such as the concentration of the proteins and the shear rate. For perfusion flow experiments, the investigators need fresh whole blood because platelets are viable for four hours. After this time, new blood is needed.

Study population: For this study the investigators need blood from human volunteers with a coagulation defect in one of the proteins of the contact activation system, e.g. FXII, FXI, prekallikrein or HMWK and controls without any coagulation defects.

Main study parameters/endpoints: The investigators main study endpoint is the ex vivo formation of platelet-mediated thrombi on collagen in a perfusion flow model. The investigators hypothesize that thrombi formed from blood of patients deficient in FXII or FXI are less stable than those formed from blood from controls.

ELIGIBILITY:
Inclusion Criteria:

* Patient group:
* Age: ≥ 18 years
* Deficiency in factor XII, factor XI, prekallikrein or high molecular weight kininogen
* Control group:
* Age: ≥ 18 years

Exclusion Criteria:

* (Other) Coagulation defects
* Symptoms of active disease
* The use of antiplatelet drugs
* The use of aspirin/ascal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients:
  Patients with a congenital factor XII-deficiency Patients with a congenital factor XI-deficiency Patients with a congenital prekallikrein-deficiency Patients with a congenital high molecular weight kininogen-deficiency
  Controls:
  Healthy individuals without any coagulation defects
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2011-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Thrombus formation, stability and break down | Up to 36 months
  Using perfusion-flow experiments the formation, stability and break down of clots formed from the blood of the study participants will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Ten Cate, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands